CLINICAL TRIAL: NCT05776394
Title: Study on Hypertension and Frailty in the Older People: the HYPER-FRAIL Study
Brief Title: Study on Hypertension and Frailty in the Older People
Acronym: HYPER-FRAIL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 09C214
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Frailty; High Blood Pressure
MeSH Terms: conditions — Frailty; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To estimate the linear association between daytime systolic blood pressure variability evaluated as standard deviation (SD) and frailty evaluated as Frailty index according to the Rockwood's accumulation of deficits model

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypertension according to the criteria of the European Society of Cardiology guidelines
* Consent of the patient (or legal representative) to participate in the study

Exclusion Criteria:

* Refusal of the patient or his/her legal representative
* Life expectancy of less than 6 months

Min Age: 75 Years | Sex: All
Age Groups: Older Adult
Study Population: Elderly patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Daytime systolic blood pressure variability | At baseline
  Standard deviation of daytime systolic blood pressure

SECONDARY OUTCOMES:
Nighttime systolic blood pressure variability | At baseline
  Standard deviation of nighttime systolic blood pressure
24h systolic blood pressure variability | At baseline
  Standard deviation of 24h systolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Luca, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided